CLINICAL TRIAL: NCT01700049
Title: ML28485:Phase 2B Single-site,Open-label,Nonrandomized Study Evaluating Efficacy of Oral Vismodegib in Various Histologic Subtypes (Infiltrative/Morpheaform,Nodular and Superficial)of High Risk and/or Locally Advanced Basal Cell Carcinoma
Brief Title: Study Evaluating the Efficacy of Oral Vismodegib in Various Histologic Subtypes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Scott W. Fosko, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28485; 22355 (Other: Saint Louis University)
Record Dates: First submitted 2012-09-25; First posted 2012-10-04 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Basal Cell Carcinoma
Keywords: advanced BCC; high risk; locally advanced
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label oral vismodegib (Experimental): This is a Phase 2B single-site, open-label, nonrandomized 24-week study of the efficacy and safety of vismodegib (150 mg PO daily) in subjects with high risk and/or locally advanced basal cell carcinoma (BCC). A total of 36 subjects with infiltrative/morpheaform, nodular, or superficial BCC will be enrolled in the study.
  Interventions: Drug: vismodegib (150 mg PO daily)

INTERVENTIONS:
Drug: vismodegib (150 mg PO daily) — Biopsies will be performed on all participants at baseline, week 12 and week 24.
  Other Names: Brand name: Erivedge

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of oral vismodegib therapy in the treatment of different 'histologic subtypes' of basal cell skin cancer (BCC). The term 'histologic subtype' refers to how the cells and tumor tissue looks under the microscope. Three different 'histologic subtypes' of basal cell skin cancer (infiltrative/morpheaform, nodular and superficial) will be examined in this study.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety and effectiveness of oral vismodegib therapy in the treatment of different 'histologic subtypes' of basal cell skin cancer (BCC). The term 'histologic subtype' refers to how the cells and tumor tissue looks under the microscope. Three different 'histologic subtypes' of basal cell skin cancer (infiltrative/morpheaform, nodular and superficial) will be examined in this study. Each subtype has a characteristic look under the microscope, which is related to how the tumor will behave and grow.

ERIVEDGE (oral vismodegib capsule) has been approved for use in the United States for treatment of metastatic BCC tumors (mBCC), tumors that have spread further into the skin, bones or other tissues, or spread to other parts of the body and locally advanced basal cell skin cancer (laBCC), cancers that have come back after surgery or that the healthcare provider thinks cannot be treated with surgery or radiation. It works by blocking the signal, called Hedgehog, which basal cell skin cancer cells need to grow. It has been given to about 800 people during clinical trials.

Data from previous studies is mostly based on a subtype of BCC made up of little round collections of cancer cells, called "Nodular". There is almost no data on the use of vismodegib in other subtypes of BCC that that tend to extend deep into the skin ("Infiltrative" subtype), or spread widely near the surface of the skin ("Superficial" subtype).

A total of 36 subjects will be enrolled in the study. All study participants will receive oral vismodegib treatment.

At the Week 12 visit, skin biopsies will be performed to give the investigators more information on how the tumor is responding to vismodegib. If there is no evidence of tumor on the biopsy, the subject will be eligible to end treatment early and enter the Observation period. During this time the subject will be followed clinically every 3 months for up to 1 year.

For all other subjects, if any evidence of tumor is seen on biopsy at week 12, the subject will continue treatment for the full 24 weeks. At week 24 visit, skin biopsies will be performed again to see if there is any tumor left. If there is no evidence of tumor on the biopsy, the subject will be eligible to end treatment early and enter the Observation period. If there is tumor left, the subject will be referred for surgery or other standard of care treatment to remove the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and data informed consent
2. Willing to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
3. 18 years of age or older at time of informed consent
4. Have one or more clinically suspicious lesions for BCC at Pre-Study screening Visit that has:

   1. a diameter ≥ 6 mm if located on the "mask areas" of face (central face, eyelids, eyebrows, periorbital,nose,lips,chin,mandible,preauricular and postauricular skin/sulci,temple,ear),genitalia,hands,or feet
   2. a diameter ≥ 10 mm if located on cheeks,forehead,scalp,or neck
   3. a diameter ≥ 20 mm if located on trunk and extremities

      or has a lesion suspicious for locally advanced BCC defined as a lesion that:
   4. is ≥ 10 mm,
   5. has recurred following surgery or surgical resection would result in substantial deformity, and
   6. has been deemed not appropriate for radiation.
5. Have a histologically-confirmed BCC prior to first dose of study drug
6. Have an Eastern Cooperative Oncology Group performance status of 2 or less at Baseline
7. Female of reproductive potential must use 2 effective methods to avoid pregnancy during therapy and for 7 months after completing therapy
8. Male patients must use effective measures to avoid pregnancy in their partner at all times during treatment and for 2 months after the last dose
9. Agree not to donate blood or blood products during the study and for 7 months after the last dose
10. Subjects with Basal Cell Nevus Syndrome are eligible for enrollment

Exclusion Criteria:

1. Women who are pregnant, lactating, or planning pregnancy while in the study
2. History of prior treatment with vismodegib or any Hh Pathway Inhibitor
3. Evidence of clinically significant and unstable diseases or conditions; Subjects with clinically stable chronic medical conditions will be allowed to enter the study
4. Any dermatological disease at treatment site that the investigator thinks may be exacerbated by treatment with vismodegib or cause difficulty with examination
5. The target lesion identified at Pre-study Screening visit has been determined to be mBCC by radiological assessment prior to first dose of study drug
6. Inability or unwillingness to swallow capsules
7. History of infection requiring hospitalization, IV antimicrobial therapy, or is otherwise judged to be clinically significant by the investigator within 4 wks prior to first dose of study drug
8. History of infection requiring antimicrobial therapy within 2 wks prior to first dose of study drug
9. History of alcohol or substance abuse, unless in full remission for greater than 6 months prior to first dose of study drug
10. Known to be infected with human immunodeficiency virus, hepatitis B or hepatitis C viruses
11. Participation in other study using an investigational or experimental therapy or procedure within 4 weeks or 5 half-lives (whichever is longer) before the study begins and/or during study participation
12. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results in the judgment of the investigator
13. Subjects who are study site staff members or who are Sponsor employees directly involved in the conduct of the trial
14. A subject who, in the opinion of the investigator or sponsor, will be uncooperative or unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2018-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Fosko, MD, Study Director — fosko.scott@mayo.edu
Locations (1):
- Saint Louis University Department of Dermatology, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorusso PM, Jimeno A, Dy G, Adjei A, Berlin J, Leichman L, Low JA, Colburn D, Chang I, Cheeti S, Jin JY, Graham RA. Pharmacokinetic dose-scheduling study of hedgehog pathway inhibitor vismodegib (GDC-0449) in patients with locally advanced or metastatic solid tumors. Clin Cancer Res. 2011 Sep 1;17(17):5774-82. doi: 10.1158/1078-0432.CCR-11-0972. Epub 2011 Jul 13. PMID 21753154
- [Background] Walling HW, Fosko SW, Geraminejad PA, Whitaker DC, Arpey CJ. Aggressive basal cell carcinoma: presentation, pathogenesis, and management. Cancer Metastasis Rev. 2004 Aug-Dec;23(3-4):389-402. doi: 10.1023/B:CANC.0000031775.04618.30. PMID 15197337
- [Background] Sekulic A, Migden MR, Oro AE, Dirix L, Lewis KD, Hainsworth JD, Solomon JA, Yoo S, Arron ST, Friedlander PA, Marmur E, Rudin CM, Chang AL, Low JA, Mackey HM, Yauch RL, Graham RA, Reddy JC, Hauschild A. Efficacy and safety of vismodegib in advanced basal-cell carcinoma. N Engl J Med. 2012 Jun 7;366(23):2171-9. doi: 10.1056/NEJMoa1113713. PMID 22670903
- [Background] Tang JY, Mackay-Wiggan JM, Aszterbaum M, Yauch RL, Lindgren J, Chang K, Coppola C, Chanana AM, Marji J, Bickers DR, Epstein EH Jr. Inhibiting the hedgehog pathway in patients with the basal-cell nevus syndrome. N Engl J Med. 2012 Jun 7;366(23):2180-8. doi: 10.1056/NEJMoa1113538. PMID 22670904
- [Background] Von Hoff DD, LoRusso PM, Rudin CM, Reddy JC, Yauch RL, Tibes R, Weiss GJ, Borad MJ, Hann CL, Brahmer JR, Mackey HM, Lum BL, Darbonne WC, Marsters JC Jr, de Sauvage FJ, Low JA. Inhibition of the hedgehog pathway in advanced basal-cell carcinoma. N Engl J Med. 2009 Sep 17;361(12):1164-72. doi: 10.1056/NEJMoa0905360. Epub 2009 Sep 2. PMID 19726763
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Oral Vismodegib: This is a Phase 2B single-site, open-label, nonrandomized 24-week study of the efficacy and safety of vismodegib (150 mg PO daily) in subjects with high risk and/or locally advanced basal cell carcinoma (BCC).
  vismodegib (150 mg PO daily): Biopsies will be performed on all participants at baseline, week 12 and week 24.
Period: Overall Study
Arm/Group | Open Label Oral Vismodegib
Started | 28
Completed | 27
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label Oral Vismodegib: This is a Phase 2B single-site, open-label, nonrandomized 24-week study of the efficacy and safety of vismodegib (150 mg PO daily) in subjects with high risk and/or locally advanced basal cell carcinoma.
  vismodegib (150 mg PO daily): Biopsies will be performed on all participants at baseline, week 12 and week 24.
Arm/Group | Open Label Oral Vismodegib
Number analyzed (Participants) | 28
Age, Continuous [Median (Standard Deviation); unit: years] | 69.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Vismodegib
Description: The efficacy of vismodegib was defined as the number of tumor biopsies with positive pathology after 24 weeks. Subjects had one target lesion and up to 3 additional non-target lesions. A cumulative total of 65 tumors was measured after 24 weeks of treatment. Histopathological subtypes were categorized primarily as infiltrative, nodular and superficial.
Time Frame: Week 24
Population: A total of 65 tumors were categorized into histopathologic subtype where 24 of 65 were infiltrative, 29 of 65 were nodular, 10 of 65 were superficial and 2 out of 65 were keratotic.
Measure: Count of Units; unit: tumors
Units Other Than Participants: tumors
Arm/Group | Open Label Oral Vismodegib
Number analyzed (Participants) | 27
Number analyzed (tumors) | 65
tumors
  Infiltrative: number analyzed (tumors) | 24
  Infiltrative | 2
  Nodular: number analyzed (tumors) | 29
  Nodular | 5
  Superficial: number analyzed (tumors) | 10
  Superficial | 1
  Keratotic: number analyzed (tumors) | 2
  Keratotic | 1

2. Secondary Outcome: Safety of Vismodegib
Description: The safety of Vismodegib was evaluated by monitoring adverse effects. All adverse events, expected and unexpected, were recorded and categorized using the Common Terminology Criteria for Adverse Events (CTCAE) guide. This is a set of criteria from the National Cancer Institute (NCI) used to standardize classification of adverse effects of drugs. Grade 1 events are defined as mild, grade 2 as moderate, grade 3 as severe; grade 4 as life-threatening and grade 5 as death.
Time Frame: Up to 18 months
Measure: Number; unit: adverse events
Arm/Group | Open Label Oral Vismodegib
Number analyzed (Participants) | 28
adverse events
  Grade 1 | 133
  Grade 2 | 48
  Grade 3 | 8
  Grade 4 | 1
  Grade 5 | 2

3. Secondary Outcome: Onset of Efficacy of Vismodegib
Description: Onset of efficacy was measured by tumor surface area reduction or increase. Subjects had one target lesion and up to 3 additional non-target lesions. Surface area of a cumulative total of 65 tumors (27 target lesions and 38 non-target lesions) was measured after 24 weeks of treatment. A complete response was defined as 100% reduction in tumor surface area. Partial response was defined as greater than 50% reduction in tumor surface area. Stable disease was defined as less than 50% reduction in tumor surface area and Progressive disease was defined as greater than 20% increase in tumor surface area.
Time Frame: Up to week 24
Measure: Count of Units; unit: tumors
Units Other Than Participants: tumors
Arm/Group | Open Label Oral Vismodegib
Number analyzed (Participants) | 27
Number analyzed (tumors) | 65
tumors
  Complete response | 13
  Partial response | 27
  Stable Disease | 24
  Progressive Disease | 1

ADVERSE EVENTS:
Time Frame: The study period during which all Adverse Events (AE) and Serious Adverse Events (SAE) must be reported begins after informed consent is obtained and initiation of study treatment and ends 30 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier.
Arm/Group | Open Label Oral Vismodegib
All-Cause Mortality (participants affected / at risk) | 2/28
Serious Adverse Events (participants affected / at risk) | 4/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Oral Vismodegib (N=28)
Myocardial infarction (Cardiac disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Neurogenic claudication (Nervous system disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Exacerbation of low back pain (General disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Oral Vismodegib (N=28)
Dysgeusia/Loss of Taste (General disorders) | 24 (24)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 23 (23)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (20)
Decreased appetite/anorexia/weight loss (Metabolism and nutrition disorders) | 9 (9)
Nausea (General disorders) | 8 (8)
Fatigue (General disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Joint aches (Musculoskeletal and connective tissue disorders) | 5 (5)
Upper respiratory infection (Infections and infestations) | 5 (5)
Itching/pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Swelling (General disorders) | 4 (4)
Muscle aches (Musculoskeletal and connective tissue disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Wound infection (Infections and infestations) | 2 (2)
Abnormal hair growth (General disorders) | 2 (2)
Insomnia (General disorders) | 2 (2)
Comedones (Skin and subcutaneous tissue disorders) | 2 (2)
Scalp tenderness (General disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Headache (General disorders) | 2 (2)
Blurry vision (Eye disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Falls (General disorders) | 2 (2)
Vomiting (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Decrease in eyelashes/eyebrows (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Biopsy site inflammation (Skin and subcutaneous tissue disorders) | 1 (1)
Viral syndrome (Infections and infestations) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Stunted nail growth (General disorders) | 1 (1)
Maxillary fibrous cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (General disorders) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1)
Dry mouth (General disorders) | 1 (1)
Tooth pain (General disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Numbness (General disorders) | 1 (1)
Rhinorrhea (General disorders) | 1 (1)
Rosacea flare (Skin and subcutaneous tissue disorders) | 1 (1)
Visual hallucinations (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Dislocation (Musculoskeletal and connective tissue disorders) | 1 (1)
Sprain (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning sensation of tongue (General disorders) | 1 (1)
Halitosis (General disorders) | 1 (1)
Eyelid reconstruction (Surgical and medical procedures) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Peripheral arterial disease (Vascular disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Sinus infection (Infections and infestations) | 1 (1)
Salivary gland infection (Infections and infestations) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Orthostatic tremor (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower extremity edema/intermittent swelling (General disorders) | 1 (1)
Elevated blood pressure (Cardiac disorders) | 1 (1)
Squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Vitamin D deficiency (General disorders) | 1 (1)
Hyperlipidemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT01700049/Prot_SAP_000.pdf